CLINICAL TRIAL: NCT02400528
Title: Prospective Cohort Follow-up of French Patients With Profound and Multiple Disabilities: Healthcare Pathways and Quality of Life Among Patients and Their Families
Acronym: Eval-PLH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-21; RCAPHM14_0082 (Other: APHM); 2014-A00953-44 (Other: IDRCB ANSM)
Record Dates: First submitted 2015-02-04; First posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-02

CONDITIONS: Paraparesis; Tetraparesis; Hemiparesis; Ataxia; Neuromuscular Disorders; Extrapyramidal Motor Disorders
MeSH Terms: conditions — Paraparesis; Quadriplegia; Paresis; Ataxia; Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients With Profound and Multiple Disabilities (Other)
  Interventions: Behavioral: quality of life questionnaires

INTERVENTIONS:
Behavioral: quality of life questionnaires

SUMMARY:
The studies conducted so far concerning the medical and paramedical cares provided to patients with profound and multiple disabilities (PMD) often show important limitations: samples are too small or very heterogeneous, generally constituted of children only; studies are mainly cross-sectional and retrospective, focusing on very specific issues instead of assessing health and quality of life from a more global perspective… So far, the investigators found no published data from a prospective cohort study involving a representative sample of patients with PMD. The present project aims to set up such a cohort so as to describe for the first time the natural history of French patients with PMD as well as the cares they receive at home or within the different dedicated structures in France. This cohort will also make it possible to identify the factors responsible for differences in the cares patients are provided, the consequences of these differences on their health and their quality of life (and those of their relatives) as well as the evolutions of these data over time. It will then allow for assessing the effectiveness of the French healthcare system to care for patients with PMD as well as building a frame of reference regarding the best cares to provide to these patients.

The primary goal of this study is to identify the determinants of health among patients with PMD.

ELIGIBILITY:
Inclusion Criteria:

* age > 3 years old,
* patient with health insurance,
* causal brain injury before the age of 3,
* Intellectual Quotient < 40 or not assessable,
* motor disability: paraparesis, tetraparesis, hemiparesis, ataxia, neuromuscular disorders, or extrapyramidal motor disorders,
* score at the Gross Motor Function Classification System > 3,
* score at the Functional Independence Measure < 55.

Exclusion Criteria:

Subject declaring benefit "psychotropic treatment which" significantly alter the reasoning, discernment or judgment.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Caregivers quality of life | 36 months
  Assessment of quality of life from questionnaires,WHOQOL-Bref, Brief-COPE
  - Brief-COPE

SECONDARY OUTCOMES:
emotional distress and subjective burden of natural caregivers, | 36 months
  Assessment of quality of life from questionnaires,WHOQOL-Bref
  * Brief-COPE
  * CRA
burnout of institutional caregivers | 36 months
  Assessment of quality of life from questionnaires,WHOQOL-Bref
  * Brief-COPE
  * MBI

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Baumstarck K, Del Duca S, El Ouazzani H, Hamouda I, Beltran Anzola A, Aim MA, Rousseau MC. Increased Life Expectancy of People With Profound Intellectual and Multiple Disabilities: What Does It Change for Parents? J Appl Res Intellect Disabil. 2025 Jan;38(1):e70018. doi: 10.1111/jar.70018. PMID 39934966
- [Derived] Rousseau MC, Beltran A, Hamouda I, Aim MA, Felce A, Lind K, Khaldi N, El Ouazzani H, Auquier P, de Villemeur TB, Baumstarck K. Impact of caring for patients with polyhandicap on institutional health care workers' quality of life: a cross-sectional and longitudinal evaluation. Front Public Health. 2024 Oct 18;12:1427289. doi: 10.3389/fpubh.2024.1427289. eCollection 2024. PMID 39494083
- [Derived] Baumstarck K, Hamouda I, Aim MA, Anzola AB, Khaldi-Cherif S, Felce A, Maincent K, Lind K, Auquier P, Billette de Villemeur T, Rousseau MC; and the EVAL-P. L. H. Group. Health care management adequacy among French persons with severe profound intellectual and multiple disabilities: a longitudinal study. BMC Health Serv Res. 2024 Jan 18;24(1):99. doi: 10.1186/s12913-024-10552-9. PMID 38238747
- [Derived] Hamouda I, Rousseau MC, Beltran Anzola A, Aim MA, de Villemeur TB, Auquier P, Baumstarck K; EVAL-PLH group. The French EVAL-PLH cohort of persons with polyhandicap. Sci Rep. 2022 Jul 22;12(1):12512. doi: 10.1038/s41598-022-16596-3. PMID 35869128
- [Derived] Rousseau MC, Baumstarck K, Valkov M, Felce A, Brisse C, Khaldi-Cherif S, Loundou A, Auquier P, Billette de Villemeur T; French Polyhandicap Group. Impact of severe polyhandicap cared for at home on French informal caregivers' burden: a cross-sectional study. BMJ Open. 2020 Feb 2;10(1):e032257. doi: 10.1136/bmjopen-2019-032257. PMID 32014871
- [Derived] Rousseau MC, Billette de Villemeur T, Khaldi-Cherif S, Brisse C, Felce A, Baumstarck K, Auquier P; French Polyhandicap Group. Adequacy of care management of patients with polyhandicap in the French health system: A study of 782 patients. PLoS One. 2018 Jul 6;13(7):e0199986. doi: 10.1371/journal.pone.0199986. eCollection 2018. PMID 29979745